CLINICAL TRIAL: NCT03133689
Title: Alcohol Consumption and Time-to-onset for Coronary Heart Disease: An Individual Participant Data Meta-analysis
Brief Title: Alcohol Consumption and Coronary Heart Disease Onset
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); Alcohol Research UK (Other)
Responsible Party: Sponsor
Other Study IDs: UCLAlcoholLifecourse_CHDStudy
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-04

CONDITIONS: Coronary Heart Disease
Keywords: Alcohol; Coronary heart disease; Ischemic heart disease; Cardiovascular health; Individual participant data meta-analysis; Longitudinal
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- EPIC-Norfolk: This cohort comprises 25,636 residents of a predefined English healthcare region (11,606 men and 14,030 women). Participants in this cohort study were originally recruited from 35 general practices in Norfolk, England as part of an investigation into diet and cancer, but the study's scope was subsequently widened to include additional outcomes including cardiovascular diseases.
- GAZEL: This cohort comprises 20,625 employees of French gas and electricity companies (15,011 men and 5,614 women). The cohort commenced data collection in 1989 and follow-up assessments were subsequently completed on an annual basis. The data have undergone linkage to national health administrative datasets.
- NSHD: This dataset comes from the 1946 National Birth Cohort study, which comprises all persons born in England, Scotland and Wales in one week in March 1946. The cohort comprises 5,362 individuals (2,815 men and 2,547 women). Data have been collected from participants on a regular basis throughout their life, including information on lifestyle and, in combination with administrative datasets, on health outcomes.
- Twenty-07-1930s: This cohort comprises 1,551 Scottish participants (702 men and 849 women) born around 1932 who were recruited in 1986 as part of a study of health inequalities. The repeated nature of the data collection will enable identification of longitudinal alcohol intake patterns, while linkage to Scottish health system records will enable identification of coronary heart disease onset.
- Twenty-07-1950s: This cohort comprises 1,444 Scottish participants (656 men and 788 women) born around 1952 who were recruited in 1986, alongside the T-07-1930s' cohort, as part of a study of health inequalities. Participant health was tracked through linkage with national health records.
- Whitehall II: This cohort comprises 10,308 British civil servants (6,895 men and 3,413 women). The cohort study commenced data collection in 1985 and participants have since undergone questionnaire and clinical assessments across regular intervals. Additional tracking of health outcomes has been performed through linkage with administrative databases. Demographic, behavioural and clinical data will be sourced from this cohort for the purposes of the current study.

SUMMARY:
The primary aim of this study is to examine if long-term patterns of alcohol consumption are associated with time-to-onset for incident coronary heart disease (fatal and non-fatal), using data from multiple cohorts.

DETAILED DESCRIPTION:
The relationship between alcohol consumption and coronary heart disease (CHD) remains an issue of debate. By capturing drinking trajectories over time, we may be equipped to obtain new insights into this relationship. Studies have shown that such trajectories have differential associations for intermediate traits (carotid intima-media thickness, pulse wave velocity and inflammatory markers), but no studies exist that link stability of drinking to actual CHD. The current study will employ a longitudinal cohort design to evaluate the association between long-term alcohol consumption trajectories and time-to-event for CHD. Data will be drawn from six cohorts (five British, one French). The combined participant pool comprises 64,926 individuals (58% male, individual cohort sizes ranging from 1,444 to 25,636 participants); those with a baseline history of CHD will be excluded. Repeat alcohol intake measurements across a 10-year interval will be the exposure, with participants' intake trajectory defined according to their alcohol consumption volume and its consistency over time. To account for heterogeneity across cohorts, individual participant data meta-analysis methods will be employed in determining CHD diagnosis rates and hazard ratios for the different intake trajectories, with adjustment for relevant demographic and clinical characteristics. Results from the modelling work illustrating the form and magnitude of the association between the alcohol intake categories and CHD will be presented.

This work will help further understanding of the role that alcohol intake and its stability over time play in subsequent CHD risk, and will have implications for our understanding of alcohol's relationship to cardiovascular health in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Participated in cohort studies being investigated
* Provided alcohol intake data at least one time point
* Was included in coronary heart disease onset tracking

Exclusion Criteria:

* Left cohort study prior to completion of 10 year exposure window
* Had history of coronary heart disease before end of 10 year exposure window

Min Age: 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be drawn from birth, regional and occupational cohort studies in England, Wales, Scotland and France.
Sampling Method: Non-Probability Sample
Enrollment: 35132 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Coronary Heart Disease | From last date of alcohol assessment until the date of hospitalisation or death due to coronary heart disease, up to 22 years depending on cohort
  Time-to-onset for coronary heart disease (fatal or non-fatal), as ascertained from linked health record data

CONTACTS AND LOCATIONS:
Overall Officials: D O'Neill, PhD, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers can request access to anonymised data. The data are already available to bona fide researchers via application: European Prospective Investigation of Cancer-Norfolk (EPIC-Norfolk; http://www.srl.cam.ac.uk/epic/contact/), Gaz et Electricité (GAZEL; http://www.gazel.inserm.fr/en/projects/submitting-a-project.html), Medical Research Council National Survey of Health and Development 1946 (NSHD; http://www.nshd.mrc.ac.uk/data/), West of Scotland Twenty-07 Study (T-07-1930s and T-07-1950s; http://2007study.sphsu.mrc.ac.uk/Information-on-data-sharing.html), and Whitehall II (WII; http://www.ucl.ac.uk/whitehallII/data-sharing).

REFERENCES:
- [Background] Britton A, Marmot MG, Shipley MJ. How does variability in alcohol consumption over time affect the relationship with mortality and coronary heart disease? Addiction. 2010 Apr;105(4):639-45. doi: 10.1111/j.1360-0443.2009.02832.x. Epub 2010 Feb 9. PMID 20148795
- [Background] Roerecke M, Rehm J. The cardioprotective association of average alcohol consumption and ischaemic heart disease: a systematic review and meta-analysis. Addiction. 2012 Jul;107(7):1246-60. doi: 10.1111/j.1360-0443.2012.03780.x. Epub 2012 Mar 21. PMID 22229788
- [Background] Marmot M, Brunner E. Cohort Profile: the Whitehall II study. Int J Epidemiol. 2005 Apr;34(2):251-6. doi: 10.1093/ije/dyh372. Epub 2004 Dec 2. No abstract available. PMID 15576467
- [Background] Day N, Oakes S, Luben R, Khaw KT, Bingham S, Welch A, Wareham N. EPIC-Norfolk: study design and characteristics of the cohort. European Prospective Investigation of Cancer. Br J Cancer. 1999 Jul;80 Suppl 1:95-103. No abstract available. PMID 10466767
- [Background] Goldberg M, Leclerc A, Zins M. Cohort Profile Update: The GAZEL Cohort Study. Int J Epidemiol. 2015 Feb;44(1):77-77g. doi: 10.1093/ije/dyu224. Epub 2014 Nov 23. PMID 25422284
- [Background] Wadsworth M, Kuh D, Richards M, Hardy R. Cohort Profile: The 1946 National Birth Cohort (MRC National Survey of Health and Development). Int J Epidemiol. 2006 Feb;35(1):49-54. doi: 10.1093/ije/dyi201. Epub 2005 Oct 4. No abstract available. PMID 16204333
- [Background] Benzeval M, Der G, Ellaway A, Hunt K, Sweeting H, West P, Macintyre S. Cohort profile: west of Scotland twenty-07 study: health in the community. Int J Epidemiol. 2009 Oct;38(5):1215-23. doi: 10.1093/ije/dyn213. Epub 2008 Oct 17. No abstract available. PMID 18930962
- [Derived] O'Neill D, Britton A, Hannah MK, Goldberg M, Kuh D, Khaw KT, Bell S. Association of longitudinal alcohol consumption trajectories with coronary heart disease: a meta-analysis of six cohort studies using individual participant data. BMC Med. 2018 Aug 22;16(1):124. doi: 10.1186/s12916-018-1123-6. PMID 30131059
- See also: University College London Research Department of Epidemiology & Public Health — https://www.ucl.ac.uk/epidemiology